CLINICAL TRIAL: NCT04052906
Title: The Effect On Self-Care and Self-Efficacy of Inhaler Training in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Gamze MUZ, Assistant Professor, Nevsehir Haci Bektas Veli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NevsehirHBVU
Record Dates: First submitted 2019-08-07; First posted 2019-08-12 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: COPD
Keywords: COPD; dyspnea; self-efficacy; self-care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Planned Inhaler Medication Training
  Interventions: Other: Training
- Control Group (No Intervention): usual care

INTERVENTIONS:
Other: Training — Planned Inhaler Medication Trainning
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the effect of planned inhaler medication training on self-care agency and self-efficacy level.

DETAILED DESCRIPTION:
Pulmonary diseases are a major source of mortality and morbidity globally. The major symptom of COPD is dyspnea. Since dyspnea leads to activity limitation and inadequate self-care skills among individuals, it is often associated with major psychological comorbidity, social isolation and poor perceived quality of life. COPD patients with high self-efficacy are high enough to level of treatment adherence. On the other hand, the most preferred treatment method for the management and mitigation of COPD symptoms is by the use of inhaler medication. However, incorrect use of the inhaler would lead to failure in the control of COPD patients. Also, it fails to provide COPD patients with self-care agency and self-efficacy levels. In COPD, planned inhaler medication training has been shown in many studies to reduce dyspnoea, increase self-care and self-efficacy levels. Therefore, planned inhaler medication training increases quality of life in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are literate,
* Diagnosed with COPD at least six months ago,
* Using inhaler medication since three or more months,
* Moderate or severe COPD, according to GOLD criteria,
* Incorrect use inhaler medication uses according to the list of inhaler medication use skills,
* No communication problems,
* No mental confusion or any psychiatric problem,
* Agrees to participate in the study.

Exclusion Criteria:

* Cognitive dysfunction,
* Severe pulmonary, cardiological or malignant disease,
* In a period of exacerbation,
* Correctly performs all steps for their prescribed inhaler medication(s), according to the list of inhaler skills.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
COPD Self-Efficacy Scale (CSES) | baseline to the 3 months after intervention
  CSES developed by Wigal et al. (1991) is used to determine the degree of confidence that COPD patients have in managing or avoiding breathing difficulty during certain activities. The scale consists of 34 items and 5 subscales.
Self-Care Agency Scale | baseline to the 3 months after intervention
  The Self-care Agency Scale (1979) was developed by Kearney and Fleischer, and its validity and reliability study in Turkey was conducted by Nahcivan in 1993. With this scale consisting of 35 items, patients evaluate their ability or agency to perform self-care actions.

SECONDARY OUTCOMES:
Modified Borg Dyspnea Scale | baseline to the 3 months after intervention
  While the Modified Borg Scale is nowadays generally used to define the severity of dyspnea in exercise, it can also be used to assess the severity of resting dyspnea
Medical Research Council (MRC) Dyspnea Scale | baseline to the 3 months after intervention
  The dyspnea scale is a 1 to 5 score scale consisting of five items based on various physical activities that produce a feeling of dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Muz, PhD, Study Chair — Nevsehir Haci Bektas Veli University
Locations (1):
- Gamze Muz, Nevşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kearney BY, Fleischer BJ. Development of an instrument to measure exercise of self-care agency. Res Nurs Health. 1979 Mar;2(1):25-34. doi: 10.1002/nur.4770020105. No abstract available. PMID 254279
- [Background] Wigal JK, Creer TL, Kotses H. The COPD Self-Efficacy Scale. Chest. 1991 May;99(5):1193-6. doi: 10.1378/chest.99.5.1193. PMID 2019177
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] FLETCHER CM. The clinical diagnosis of pulmonary emphysema; an experimental study. Proc R Soc Med. 1952 Sep;45(9):577-84. No abstract available. PMID 13003946
- [Result] Goris S, Tasci S, Elmali F. The effects of training on inhaler technique and quality of life in patients with COPD. J Aerosol Med Pulm Drug Deliv. 2013 Dec;26(6):336-44. doi: 10.1089/jamp.2012.1017. Epub 2013 Feb 19. PMID 23421900